CLINICAL TRIAL: NCT01528306
Title: An Exploratory, Cross-Over Study of the Safety of HP802-247 Applied to Open Wounds of Subjects With Dystrophic Epidermolysis Bullosa
Brief Title: A Pilot Study of HP802-247 in Dystrophic Epidermolysis Bullosa
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802-247-09-026
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: HP802-247; EB (epidermolysis bullosa)
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HP802-247 (Experimental)
  Interventions: Biological: HP802-247
- Placebo (Vehicle) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HP802-247 — Wounds up to 12 cm2: 1 spray each component (0.5 x 106 cells per mL allogeneic human keratinocytes and fibroblasts) applied weekly as a topical spray for up to 4 weeks in each of 2 treatment periods
  Larger wounds:
  (>12 cm2 and ≤ 24 cm2) 2 sprays each; (>24 cm2 and ≤ 36 cm2) 3 sprays each; (>36 cm2 and ≤ 48 cm2) 4 sprays each
  Arms: HP802-247
Other: Placebo — Wounds up to 12 cm2: 1 spray each component (thrombin solution and fibrinogen solution) applied weekly as a topical spray for up to 4 weeks in each of 2 treatment periods
  Larger wounds:
  (>12 cm2 and ≤ 24 cm2) 2 sprays each; (>24 cm2 and ≤ 36 cm2) 3 sprays each; (>36 cm2 and ≤ 48 cm2) 4 sprays each
  Arms: Placebo (Vehicle)

SUMMARY:
This is a pilot study designed to see if HP802-247, an investigational treatment with living human skin cells, helps to heal blisters or wounds in subjects with Dystrophic Epidermolysis Bullosa (DEB). The durability of the skin in healed wounds treated with HP802-247 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written consent must be obtained from a parent or legally authorized representative. Assent will be obtained according to local requirements.
* Subjects with a clinical diagnosis of DEB with recurring blisters, ≥ 2 years of age at Screening. Subjects may be of either sex and of any race or skin type provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* A parent or legally authorized representative must be willing and able to ensure subject is present for all required study visits.
* A parent or legally authorized representative must be able to follow instructions.
* Have an open wound for ≤ 72 hours that:

  * is still open and has not scabbed or crusted over
  * has no dermatologic disease and/or condition in the treatment area (other than DEB with recurring blisters), including active or recent infection (within 7 days) that may be exacerbated by treatment, require treatment with antibiotics / antifungals /antivirals, require a surgical intervention, or cause difficulty with examination
  * is ≥ 4 cm² and ≤ 48 cm2 in total area (open portion)
* Females of childbearing potential (defined as post-menarcheal as documented in the medical history) may participate in the study if they meet all of the following conditions:

  * they are not breast feeding;
  * they have a negative urine pregnancy test at Week 1 Period 1;
  * they agree to undertake scheduled urine pregnancy tests at Week 1 for Periods 1, 2, & 3 and at study exit
  * they do not intend to become pregnant during the study;
  * they are using adequate birth control methods and they agree to continue using those methods for the duration of the study
* A parent or legally authorized representative must be willing and able to ensure subject is present for all required study visits (for minor subjects)
* A parent or legally authorized representative must be able to follow instructions (for minor subjects)

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the test article, their components (e.g., aprotinin, fibrinogen), or substances used in the manufacture of the test article (e.g., penicillin, streptomycin, amphotericin B, bovine serum albumin).
* Therapy with another investigational agent within thirty (30) days of the Screening Visit, or during the study.
* Have uncontrolled intercurrent or chronic illness that, in the opinion of the Investigator, would limit compliance with study requirements, represents a potential safety risk, or require treatment with an excluded drug/treatment.
* The Investigator or Medical Monitor may declare any subject ineligible for a valid medical reason.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Time to healing | 4 weeks
  Time to healing, defined as the number of days between wound onset (caregiver reported) and complete epithelialization (Investigator assessed).

SECONDARY OUTCOMES:
Wound pain as measured by faces pain scale | 4 weeks for each of 3 treatment periods
  Change from baseline (i.e., Week 1 of each period) in wound pain for each visit (Weeks 2-5 of each treatment period)as assessed by the Faces Pain Scale (FPS)
Percent of change in wound area | 4 weeks for each of 3 treatment periods
  Percent of change from baseline (i.e., Week 1 of each period) in the target wound area for each visit and Weeks 2-5 of each treatment period.
Persistence of healing | 4 weeks for each of 3 treatment periods
  Persistence of healing as assessed by lack of blister/wound recurrence for healed wounds of each period (up to 40 weeks following enrollment)
Burning and stinging upon application | 4 weeks for each of 3 treatment periods
  Burning and stinging upon application of HP802-247 or its Vehicle will be assessed at each visit of each period with the exception of the end of treatment visit (Weeks 1-4 of treatment period).
  Burning/stinging scale is a four point scale (i.e., none, mild, moderate, severe).

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Jaime E Dickerson, PhD, Study Director — Healthpoint; Herbert B Slade, MD, Principal Investigator — Healthpoint